CLINICAL TRIAL: NCT05195840
Title: A Pilot Investigation of Network-Informed Personalized Treatment for Eating Disorders Versus Enhanced Cognitive Behavioral Therapy and Dynamic Mechanisms of Change
Brief Title: Personalized Treatment for Eating Disorders Versus CBT-E Trial
Acronym: PT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Cheri Levinson, Associate Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#: 21.0689; 3R34MH128213-01S1 (NIH)
Record Dates: First submitted 2022-01-04; First posted 2022-01-19 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Eating Disorders
Keywords: eating disorder; treatment; anorexia nervosa; bulimia nervosa; binge eating disorder; atypical anorexia nervosa; therapy; other specified feeding and eating disorder
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized Treatment for Eating Disorders (Experimental): Participants will complete 3 sessions of education about the treatment while completing 2 weeks of mobile application questions. After completion of treatment education and mobile application questions, participants will complete 17 sessions of personalized treatment for eating disorders.
  Interventions: Behavioral: Personalized Treatment for Eating Disorders
- Cognitive Behavioral Therapy for Eating Disorders (Active Comparator): Participants will complete 3 sessions of education about the treatment while completing 2 weeks of mobile application questions. After completion of treatment education and mobile application questions, participants will complete 17 sessions of Cognitive Behavioral Therapy for Eating Disorders.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Eating Disorders

INTERVENTIONS:
Behavioral: Personalized Treatment for Eating Disorders — The first three sessions consist of diagnosis and general psychoeducation on EDs and treatment for ED. After mobile-assessment is complete, Session 4 includes psychoeducation on the network-informed model of personalized treatment and 14 sessions (sessions 5-19) are focused on the top three targets (4-5 sessions per target). Session 20 is a termination and conclusion session.
  Arms: Personalized Treatment for Eating Disorders
Behavioral: Cognitive Behavioral Therapy for Eating Disorders — The first three sessions consist of diagnosis and general psychoeducation on EDs and treatment for ED. After mobile-assessment is complete, Session 4 consists of food monitoring, addressing irregular eating, challenging thoughts, making adaptive behavioral changes, and relapse prevention. Session 20 is a termination and conclusion session.
  Arms: Cognitive Behavioral Therapy for Eating Disorders

SUMMARY:
The scientific premise, developed from past work, is that treatment personalized based on idiographic models (termed Network Informed Personalized Treatment; NA-PT) will outperform the current gold-standard treatment (Enhanced Cognitive Behavioral Therapy: CBT-E). The study goals are to (1) develop and test the acceptability, feasibility, and preliminary efficacy of a randomization of NA-PT versus CBT-E and (2) to test if network-identified precision targets are the mechanism of change. These goals will ultimately lead to the very first personalized treatment for ED and can be extended to additional psychiatric illnesses. Specific aims are (1) To collect preliminary data on the feasibility and acceptability of the randomization of NA-PT (n=40) for EDs versus CBT-E (n=40), (2) To test the initial clinical efficacy of NA-PT versus CBT-E on clinical outcomes (e.g., ED symptoms, body mass index, quality of life) and (3) To examine if changes in NA-identified, precision targets, as well as in dynamic network structure, are associated with change in clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Meets criteria for DSM-5 defined AN, BN, BED, or OSFED (Atypical AN and Atypical BN)
* Not currently receiving psychological treatment focused on ED

Exclusion Criteria:

* Under 18
* Over 65
* Does not meet criteria for DSM-5 defined AN, BN, BED, or OSFED (Atypical AN and Atypical BN)
* High and active Suicidality
* Active Mania
* Medically Compromised Status including extremely low weight - less than or equal to 75% median BMI for age, sex, and height
* Simultaneous psychological treatment focused on ED

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Impairment using the Clinical Impairment Assessment | Up to 1-Month Follow-Up
  The Clinical Impairment Assessment (CIA), a self report measure, is assessed at multiple time points throughout the duration of the study and is used to examine the severity of psychosocial impairment caused by eating disorders. The scores range from 0 to 64 with higher scores indicating more impairment.
Change in Eating Disorder Symptoms using the Eating Disorder Examination Questionnaire | Up to 1-Month Follow-Up
  The Eating Disorder Examination Questionnaire (EDE-Q), a self report measure, is assessed at multiple time points throughout the duration of the study and is used to examine attitudes and behaviors in individuals with eating disorder symptoms. The scores range from 0-6 with higher scores indicating higher severity of eating disorder symptoms.
Change in Quality of Life using the Quality of Life Scale | Up to 1-Month Follow-Up
  The Quality of Life Scale (QOLS), a self report measure, is assessed at multiple time points throughout the duration of the study and is used to examine various domains of quality of life. Scores range from 16 to 112 with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Cheri A Levinson, PhD, Principal Investigator — University of Louisville
Locations (1):
- Eating Anxiety Treatment Laboratory and Clinic, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levinson CA, Williams BM. Eating disorder fear networks: Identification of central eating disorder fears. Int J Eat Disord. 2020 Dec;53(12):1960-1973. doi: 10.1002/eat.23382. Epub 2020 Sep 12. PMID 32918319
- [Background] Levinson CA, Vanzhula I, Brosof LC. Longitudinal and personalized networks of eating disorder cognitions and behaviors: Targets for precision intervention a proof of concept study. Int J Eat Disord. 2018 Nov;51(11):1233-1243. doi: 10.1002/eat.22952. Epub 2018 Oct 6. PMID 30291641
- [Background] Murphy R, Straebler S, Cooper Z, Fairburn CG. Cognitive behavioral therapy for eating disorders. Psychiatr Clin North Am. 2010 Sep;33(3):611-27. doi: 10.1016/j.psc.2010.04.004. PMID 20599136
- [Background] Fairburn CG, Cooper Z, Shafran R. Cognitive behaviour therapy for eating disorders: a "transdiagnostic" theory and treatment. Behav Res Ther. 2003 May;41(5):509-28. doi: 10.1016/s0005-7967(02)00088-8. PMID 12711261